CLINICAL TRIAL: NCT05757518
Title: Cryosauna for Post-exercise Recovery of Delayed Onset Muscle Soreness (DOMS) in Recreational Athletes: a Randomized Control Trial
Brief Title: Post-exercise Recovery of DOMS in Recreational Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wroclaw University of Health and Sport Sciences (Other)
Collaborators: Gdansk University of Physical Education and Sport (Other)
Responsible Party: Principal Investigator, Sebastian Klich, Study Director, Wroclaw University of Health and Sport Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: AWFiS#1/2023; KB-62/22 (Other: Regional Medical Society in Gdynia)
Record Dates: First submitted 2023-02-11; First posted 2023-03-07 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Injury;Sports
Keywords: DOMS; injury prevention; performance; muscle properties
MeSH Terms: conditions — Athletic Injuries

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants will be allocated to intervention (cryostimulation using cryosauna) or a control group (without any intervention) using a randomized list of allocated numbers generated by a computer program. The investigator and Outcomes Assessor will be blinded to the allocation process.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Cryo-stimulation using cryosauna after fatigue-induced exercise.
  Interventions: Other: Cryosauna
- Control group (No Intervention): Without any intervention after fatigue-induced exercise.

INTERVENTIONS:
Other: Cryosauna — The intervention was Cryosauna - cryostimulation at -110°C for 1.5 minutes, for four consecutive days.
  Arms: Experimental group

SUMMARY:
The main goal of this study was to investigate the effectiveness of cryo-sauna in preventing the development of DOMS in the lower extremity. The second goal is to analyze the rate of regenerative changes in the right muscles after acute fatigue-induced exercises.

DETAILED DESCRIPTION:
The main goal of this study was to investigate the effectiveness of cryo-sauna in preventing the development of DOMS in the lower extremity. The second goal is to analyze the rate of regenerative changes in the right muscles after acute fatigue-induced exercises.

This study design was a randomized, controlled single-blind trial with repeated measures. Moreover, the design was prepared according to the Consolidated Standards of Reporting Trials (CONSORT) for pragmatic trials. Participants were assigned into two groups: (1) experimental group (CRYO, n =16) - cryostimulation using a cryo sauna; and (2) control group (CONT, n = 15) - without any intervention. This study was conducted in the Physical Exercise Laboratory. Both groups, CRYO and CON performed a fatigue-induced protocol consisting of counter-movement jumps (CMJ) (10 set for 10 repetitions). After the fatigue exercises, only CRYO underwent cryo sauna intervention including entry immediately after, 24, 48, and 72 hours post-exercise. The order of measurements at baseline included: blood sample testing (creatine kinase, myoglobin, leukocytes) and muscle stiffness of the lower extremity. All measurements we collected at baseline, immediately post, 24, 48, 72, and 96 hours post-exercise.

ELIGIBILITY:
Inclusion Criteria:

* no previous experience with cryostimulation using a cryo-sauna,
* recreational lifestyle.

Exclusion Criteria:

* Current or prior pain or injury in the lower extremity.
* Previous history of surgery in the lower extremity.
* Cardiovascular disabilities.

Ages: 20 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-01-16 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Measurement of muscle stiffness in the lower extremity. | Change from baseline muscle stiffness at 96 hours after fatigue-induced exercise.
  Stiffness [N/m] was measured on: the anterior thigh, posterior thigh, shin, and calf muscles in 23 reference points.
Measurement of blood markers. | Change from baseline leukocytes concentration at 96 hours after fatigue-induced exercise.
  Leukocytes [10^9 /L] concentration.
Measurement of blood markers. | Change from baseline creatine kinase concentration at 96 hours after fatigue-induced exercise.
  Creatine kinase [ng/mL] concentration.
Measurement of blood markers. | Change from baseline myoglobin concentration at 96 hours after fatigue-induced exercise.
  Myoglobin [ng/mL] concentration.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Klich, Dr., Study Director — University School of Physical Education in Wrocław
Locations (1):
- Physical Exercise Laboratory, Gdansk, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Klich S, Krymski I, Michalik K, Kawczynski A. Effect of short-term cold-water immersion on muscle pain sensitivity in elite track cyclists. Phys Ther Sport. 2018 Jul;32:42-47. doi: 10.1016/j.ptsp.2018.04.022. Epub 2018 May 1. PMID 29738892
- [Background] Klich S, Ficek K, Krymski I, Klimek A, Kawczynski A, Madeleine P, Fernandez-de-Las-Penas C. Quadriceps and Patellar Tendon Thickness and Stiffness in Elite Track Cyclists: An Ultrasonographic and Myotonometric Evaluation. Front Physiol. 2020 Dec 14;11:607208. doi: 10.3389/fphys.2020.607208. eCollection 2020. PMID 33381054
- [Background] Kons RL, Orssatto LBDR, Sakugawa RL, da Silva Junior JN, Diefenthaeler F, Detanico D. Effects of stretch-shortening cycle fatigue protocol on lower limb asymmetry and muscle soreness in judo athletes. Sports Biomech. 2023 Sep;22(9):1079-1094. doi: 10.1080/14763141.2020.1779335. Epub 2020 Jul 9. PMID 32644009